CLINICAL TRIAL: NCT03674073
Title: A Study to Assess the Safety, Feasibility, and Immunogenicity of Personalized Neoantigen-based Dendritic Cell Vaccine in Combination With Microwave Ablation to Treat Hepatocellular Carcinoma
Brief Title: A Study Combining Personalized Neoantigen-based Dendritic Cell Vaccine With Microwave Ablation for the Treatment of Hepatocellular Carcinoma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Collaborators: Likang Life Sciences Holdings Limited (Unknown)
Responsible Party: Principal Investigator, Ping Liang, Professor, Chinese PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LKSM001
Record Dates: First submitted 2018-09-14; First posted 2018-09-17 (Actual); Last update posted 2018-10-18 (Actual); Status verified 2018-10

CONDITIONS: Hepatocellular Carcinoma; Liver Cancer, Adult
Keywords: Neoantigen; Vaccine; Dendritic Cell; Personalized; Liver cancer
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Microwave Ablation + Neoantigen Vaccines (Experimental): The HCC patients will be treated firstly by Microwave Ablation, and then treated by courses of Neoantigen Vaccines.
  Interventions: Biological: Neoantigen Vaccines; Procedure: Microwave Ablation
- Microwave Ablation (Active Comparator): The HCC patients will be treated only by Microwave Ablation.No vaccine will be used.
  Interventions: Procedure: Microwave Ablation

INTERVENTIONS:
Biological: Neoantigen Vaccines — HCC (3cm≤D ≤5 cm, fewer than three tumors) patients were treated with Microwave Ablation and 7 courses of neoantigen-based DC vaccines.The first neoantigen-based DC vaccine injection will take place up to 30 days following the completion of Microwave Ablation. The day of the first vaccine injection will be referred to as Day 1.The schedule of vaccination is Day 1, Day 8, Day 15, Day 22, Day 50, Day78, Day106.
  Other Names: Personalized Neoantigen-based Dendritic Cell Vaccine
  Arms: Microwave Ablation + Neoantigen Vaccines
Procedure: Microwave Ablation — ALL the HCC patients will be treated by Microwave Ablation.

SUMMARY:
This is a single institution, open-label, multi-arm, pilot study of a personalized neoantigen-based dendritic cell (DC) vaccine combined with microwave ablation in subjects with Hepatocellular Carcinoma (HCC). Patients with HKLC stage IIa HCC are eligible for enrollment. In this study, the investigators are looking at the safety, feasibility of the personalized neoantigen-based DC vaccine combined with microwave ablation as well as the T cell immune response to the vaccine.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed patients with primary hepatocellular carcinoma, HKLC Stage IIa.
2. Age is greater than 18 years old, male or female.
3. The tumor size is 3cm-5cm, and the lesions are <3.
4. ECOG score < 2, Child-Pugh classification A or B.
5. The participants freely sign informed consent;

Exclusion Criteria:

1. Pregnant or breast-feeding; psychiatric problems, addiction, or any other disorder that prevented informed consent;
2. Portal vein thrombosis or extrahepatic metastases;
3. White blood cell count <2 x 10e9/L, platelet count <40 x 10e9/L, serum creatinine >110 mol/L, aspartate aminotransferase >3 times upper limit, serum bilirubin > 2.5 times upper limit, prothrombin time> 19 seconds.
4. Active uncontrolled infection;
5. Concurrent systemic corticosteroid treatment
6. Primary immunodeficiency or systemic autoimmune disease; being treated with immunosuppressive drugs for other diseases;
7. Clinically significant ischemic heart disease or cardiac failure;
8. The investigator believes that there are other reasons that are not suitable for inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2018-10-15 (Estimated); Primary Completion 2020-10-15 (Estimated); Study Completion 2020-12-15 (Estimated)

PRIMARY OUTCOMES:
Safety of neoantigen-based DC vaccine as measured by the number of subjects experiencing each type of adverse event according to the National Cancer Institute Common Terminology Criteria for Adverse Events v4.0. | 1 years

SECONDARY OUTCOMES:
Immunogenicity of the neoantigen-based DC vaccine as measured by the frequency of antigen -specific T cells using ELISPOT analysis and ICS analysis. | 2 years
Number of participants alive at 2 years | 2 years
Progression-free survival at 2 years | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Ping Liang, Doctor, Principal Investigator — Chinese PLA General Hospial
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China